CLINICAL TRIAL: NCT01868256
Title: Safety of a Early Discharge Strategy in Patients With Low-risk ST-segment Elevation Myocardial Infarction Treated With Primary Coronary Intervention: a Randomized Controlled Trial
Brief Title: Safety of Early Discharge Following Low Risk Myocardial Infarction
Acronym: EDAMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-PAP-2011-07
Record Dates: First submitted 2012-11-23; First posted 2013-06-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; primary percutaneous intervention; prognosis; early discharge
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early discharge (< 72 h) (Experimental): Patients randomized the early discharge group will be discharged from the hospital in < 72 hours
  Interventions: Other: early discharge (<72 h)
- Conventional discharge (Active Comparator): Patients randomized to the conventional discharge group will be discharged according to the local hospital protocol and/or treating physician criterion
  Interventions: Other: Conventional discharge

INTERVENTIONS:
Other: early discharge (<72 h)
  Arms: Early discharge (< 72 h)
Other: Conventional discharge
  Arms: Conventional discharge

SUMMARY:
* Objectives: The primary objective of this study is to evaluate the safety of an early discharge strategy in patients with low risk ST-elevation myocardial infarction (STEMI), treated with primary percutaneous coronary intervention (PPCI), compared to a conventional strategy.
* Methodology: Unicentric, randomized, controlled, non-inferiority and open label clinical trial. The investigators will compare an early discharge strategy (≤72 hours) with a conventional strategy (discharge according to treating physician's criterion). Inclusion criteria will be: low risk (Zwolle risk score ≤3) STEMI treated with PPCI within 24 hours from symptoms onset. Exclusion criteria will be: arrhythmias (ventricular tachycardia or fibrillation, asystole, pulseless electrical activity, advanced atrio-ventricular block), mechanical complications (cardiac tamponade, free-wall or septal rupture, acute mitral regurgitation, pericarditis), severe or moderate bleeding (according to the GUSTO criteria), complications related to vascular access of the procedure, acute kidney failure, infection, heart failure. Sample size will be 1558 subjects (n=779 per group). The investigators will study demographic, clinical, biochemical, echocardiographic and angiographic variables. The primary endpoint will be a composite of death, reinfarction, new angina, heart failure, ventricular arrhythmias, stroke and severe bleeding. The secondary endpoint will include each of the items of the primary endpoint and quality of life and functional capacity questionnaire SF-36. Finally, the investigators will analyze the degree of compliance with the European Society of Cardiology guidelines on STEMI and the rate of hospitalization-related complications. Follow up will be at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* low risk (Zwolle risk score ≤3) STEMI treated with PPCI within 24 hours from symptoms onset
* Informed consent

Exclusion Criteria:

* arrhythmias (ventricular tachycardia or fibrillation, asystole, pulseless electrical activity, advanced atrio-ventricular block)
* mechanical complications (cardiac tamponade, free-wall or septal rupture, acute mitral regurgitation, pericarditis)
* severe or moderate bleeding (according to the GUSTO criteria)
* complications related to vascular access of the procedure
* acute kidney failure
* infection
* heart failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1558 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
All cause mortality, new acute myocardial infarction, new unstable angina, heart failure, ventricular arrhythmias, stroke and severe bleeding. | 1 month
  Composite primary end-point

SECONDARY OUTCOMES:
All cause mortality | 1 month
Myocardial infarction | 1 month
Unstable angina | 1 month
Heart failure | 1 month
Ventricular arrhythmias | 1 month
Stroke | 1 month
Severe bleeding | 1 month
  According to the Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO) classification

OTHER OUTCOMES:
Difference in quality of life and functional capacity questionnaire SF-36. | 1 month
Compliance of treatment | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Sionis, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Newby LK, Eisenstein EL, Califf RM, Thompson TD, Nelson CL, Peterson ED, Armstrong PW, Van de Werf F, White HD, Topol EJ, Mark DB. Cost effectiveness of early discharge after uncomplicated acute myocardial infarction. N Engl J Med. 2000 Mar 16;342(11):749-55. doi: 10.1056/NEJM200003163421101. PMID 10717009
- [Background] De Luca G, Suryapranata H, van 't Hof AW, de Boer MJ, Hoorntje JC, Dambrink JH, Gosselink AT, Ottervanger JP, Zijlstra F. Prognostic assessment of patients with acute myocardial infarction treated with primary angioplasty: implications for early discharge. Circulation. 2004 Jun 8;109(22):2737-43. doi: 10.1161/01.CIR.0000131765.73959.87. Epub 2004 May 24. PMID 15159293
- [Background] Grines CL, Marsalese DL, Brodie B, Griffin J, Donohue B, Costantini CR, Balestrini C, Stone G, Wharton T, Esente P, Spain M, Moses J, Nobuyoshi M, Ayres M, Jones D, Mason D, Sachs D, Grines LL, O'Neill W. Safety and cost-effectiveness of early discharge after primary angioplasty in low risk patients with acute myocardial infarction. PAMI-II Investigators. Primary Angioplasty in Myocardial Infarction. J Am Coll Cardiol. 1998 Apr;31(5):967-72. doi: 10.1016/s0735-1097(98)00031-x. PMID 9561995
- [Background] Kotowycz MA, Cosman TL, Tartaglia C, Afzal R, Syal RP, Natarajan MK. Safety and feasibility of early hospital discharge in ST-segment elevation myocardial infarction--a prospective and randomized trial in low-risk primary percutaneous coronary intervention patients (the Safe-Depart Trial). Am Heart J. 2010 Jan;159(1):117.e1-6. doi: 10.1016/j.ahj.2009.10.024. PMID 20102876